CLINICAL TRIAL: NCT05120531
Title: Finding the Contribution of the Autonomic Nervous System During Perioperative Events in Children With Down Syndrome
Brief Title: Down Syndrome Autonomic Nervous System Induction Bradycardia
Acronym: DANSIB
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-0643; R21HL162572 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Down Syndrome; Bradycardia
MeSH Terms: conditions — Down Syndrome; Bradycardia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Down Syndrome patients undergoing otolaryngologic surgery with anesthesia
  Interventions: Other: Monitoring patients undergoing surgery to look for association between ANS activity and bradycardia
- Non-Down Syndrome patients undergoing otolaryngologic surgery with anesthesia
  Interventions: Other: Monitoring patients undergoing surgery to look for association between ANS activity and bradycardia

INTERVENTIONS:
Other: Monitoring patients undergoing surgery to look for association between ANS activity and bradycardia — Use of an Ambulatory Monitoring System from Vuije University (VU-AMS) to record autonomic and cardiovascular activity of patients undergoing otolaryngologic surgery with anesthesia. This monitoring device will provide data of ANS activity and normoxic bradycardia among patients with Down Syndrome. This data will be compared to data from patients without Down Syndrome.

SUMMARY:
Children with Down syndrome (DS) often experience dangerously low heart rates on induction of anesthesia for routine procedures and this occurs at 10 times the rate of non-DS patients. Given that the cardiac output of children is heart rate dependent, bradycardia is especially perilous in this population.

Historically, individuals with DS were not expected to survive beyond childhood; consequently, correction of congenital anomalies, e.g. cardiac defects, was not frequently offered. Fortunately, today individuals with DS live into adulthood and surgical correction of anomalies is universally offered. Thus, increasing numbers of children with DS are exposed to anesthesia and at risk for this hemodynamic catastrophe. It is medically unacceptable and an autonomic nervous system mechanism will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are overtly healthy as determined by medical evaluation including lack of diagnosis of Down Syndrome and children with Down Syndrome

Exclusion Criteria:

1. Contraindication to adhesive placement, eg, epidermolysis bullosa
2. Patient or parent refusal
3. Opioids
4. Heart rate altering therapy such as beta blockers
5. During the study period, participants will abstain from ingesting caffeine- or xanthine-containing products (eg, coffee, tea, cola drinks, and chocolate) for [6 hours] before the start of the anesthetic.
6. Participants will be assumed not to be using tobacco or alcohol during the study period due to their young age.

Ages: 1 Month to 8 Years | Sex: All
Age Groups: Child
Study Population: The study population will be children age 1 month to 8 years undergoing otolaryngologic surgery with anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Ambulatory feasibility of VU-AMS monitor on patients with Down Syndrome | Immediately upon entry into Same Day Surgery patient room
  Subjects will be observed for monitor use coming to the hospital for surgery. The two outcomes will be binary: wearing the device or not. We anticipate that 50% of subjects will be wearing the VU-AMS monitor on entry to the hospital on the day of surgery.
Ambulatory feasibility of VU-AMS monitor on patients without Down Syndrome | Immediately upon entry into Same Day Surgery patient room
  Subjects will be observed for monitor use coming to the hospital for surgery. The two outcomes will be binary: wearing the device or not. We anticipate that 50% of subjects will be wearing the VU-AMS monitor on entry to the hospital on the day of surgery.
Operating room feasibility of VU-AMS monitor on patients with Down Syndrome | Immediately prior to mask induction with sevoflurane
  Subjects will be observed for monitor use throughout surgery. We anticipate that 80% of subjects will wear the VU-AMS in the operating room
Operating room feasibility of VU-AMS monitor on patients without Down Syndrome | Immediately prior to mask induction with sevoflurane
  Subjects will be observed for monitor use throughout surgery. We anticipate that 80% of subjects will wear the VU-AMS in the operating room
Autonomic data including pre-ejection period and respiratory sinus arrhythmia among patients with Down Syndrome | Beginning at time of bradycardia and continuing for the next 300 seconds.
  Among subjects who become bradycardic with induction of anesthesia, we expect that the pre-ejection period will increase by 20%
Autonomic data including pre-ejection period and respiratory sinus arrhythmia among patients without Down Syndrome | Beginning at time of bradycardia and continuing for the next 300 seconds.
  Among subjects who become bradycardic with induction of anesthesia, we expect that the pre-ejection period will increase by 20%

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Sinton, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States